CLINICAL TRIAL: NCT06276231
Title: Comparative Efficacy of Nebulized Salbutamol in Alleviating Acute Renal Colic Pain: A Randomized Clinical Trial
Brief Title: Nebulized Salbutamol in Acute Renal Colic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Usama Al-Khalasi, Oman Medical Specialty Board Certified Accident and Emergency Specialist, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SalbuEase
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Renal Colic
Keywords: Salbutamol
MeSH Terms: conditions — Renal Colic | interventions — Albuterol; Saline Solution; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): Patients in this group will receive the standard treatment (75mg IM Diclofenac ) + nebulized 0.9% normal saline.
  Interventions: Other: 0.9% Normal Saline; Drug: Diclofenac Injection
- Intervention Group (Experimental): Patients in this group will receive the standard treatment (75mg IM Diclofenac ) + nebulized 10 mg of Nebulized Salbutamol.
  Interventions: Drug: Salbutamol; Drug: Diclofenac Injection

INTERVENTIONS:
Drug: Salbutamol — Salbutamol 10mg nebulization over 5 minutes ( flow rate 5-7 liters).
  Other Names: Nebulized Salbutamol
  Arms: Intervention Group
Other: 0.9% Normal Saline — Normal saline nebulization over 5 minutes ( flow rate 5-7 liters).
  Other Names: Nebulized 0.9% Normal Saline
  Arms: Control Group
Drug: Diclofenac Injection — 75 mg of Diclofenac intramuscular Injection
  Other Names: Olfen 75mg IM

SUMMARY:
A Prospective, double blinded, Randomized efficacy and safety trial of Nebulized Salbutamol in acute renal colic.

Research Summary:

INTRODUCTION: Pain is a common reason for individuals to seek health care, especially emergency care. Salbutamol has an effect for smooth muscle relaxation of the ureters. The administration of Salbuatmol has been shown to be safe and effective in the treatment of asthma exacerbation, but there have been no studies evaluating the use of neublized salbutamol for the treatment of acute renal colic pain in the emergency department.

METHOD: This is a double blinded randomized clinical controlled trial. Two hundred renal colic patients presenting to the emergency department will be randomized to intervention (10 mg nebulized salbutamol) and (10 ml neublized Normal saline) case groups. Both the groups will get the standard treatment (IM diclofenac 75mg) added to the intervention. Their pain before and after intervention will be measured by Numerical Rating scale (NRS pain score). Patient and attending physician will be blinded throughout the study. The Secondry outcomes are safety, need for rescue medications and time to discharge.

AIM: The aim of this study is to compare analgesic effects of Nebulized Salbutamol versus Placebo in adult patients with renal colic.

PRIMARY OJECTIVES: Analgesic effects of Nebulized Salbutamol on the Numerical Rating scale (NRS).

SECONDARY OBJECTIVES: Adverse Events, the need of rescue pain medications and time to discharge.

PATEINT POPULATION: Adults (from age 18 to 60 years) who presents to emergency department (ED) at Armed force Hospital with acute flank pain suggestive of renal colic

INTERVENTION: Single dose of Nebulized Salbutamol 10mg.

CLINICAL MEASURMENT: Numerical pain Analog Scale will be assessed at 0,15,30, 45 and 60 minutes after intervention. Number and dosage of rescue medication, any reported events by patient or attending physician will be documented.

OUTCOME: Decrease in pain measures by NRS pain score after Nebulized Salbutamol is given, tolerability and safety evaluation.

DETAILED DESCRIPTION:
Renal colic is recognized as one of the most intense types of pain a person can experience. The occurrence of renal stones is widespread, affecting people of all ages, genders, and races, with a lifetime risk of 12%. Men, especially those between 20-49 years, are more commonly affected than women. Recent studies show an increasing number of cases in both developed and developing countries over the past years. In Oman, while renal stones are a common health issue, the exact number of cases is not known due to a lack of data. Regional research indicates a prevalence between 4-20%, with twice as many men affected as women.

The formidable impact of renal colic extends to the realm of emergency medicine, as pain ranks as the paramount driver of emergency department (ED) visits, constituting nearly 45% of all ED admissions, particularly among those grappling with moderate to severe pain. Effective pain management in this context has profound implications, fostering improved patient satisfaction, shorter hospital stays, and reduced mortality rates. Acute renal colic, characterized by its excruciating intensity, is a frequent motive for ED visits across the globe, compelling individuals to seek immediate relief. The pain in renal colic is intricately linked to the stone's location within the urinary system and may manifest concomitantly with hematuria, urinary flow obstruction, infections, or hydronephrosis.

The primary concern for individuals confronted with renal colic is the rapid alleviation of pain. The choice of analgesic hinges on a complex interplay of factors, including availability, safety, efficacy, cost considerations, and the shared preferences of both patients and healthcare providers. Within this spectrum, nonsteroidal anti-inflammatory drugs (NSAIDs) often ascend as the preferred initial choice for pain management, guided by multiple clinical practice guidelines. NSAIDs hold sway over opioids due to their superior pain relief, diminished side effect profile, and reduced demand for adjunctive painkillers.

Salbutamol, a widely employed beta-adrenoreceptor agonist, finds its niche in diverse medical conditions, distinguished by its favorable safety profile. Beta-adrenoreceptor agonists manifest a multifaceted approach to addressing the etiology of renal colic pain, countering factors such as ureteral spasms and inflammation. They exhibit the capacity to induce ureteral relaxation, mitigate muscular contractions, and alleviate renal pressure. Importantly, salbutamol's distinctive pharmacokinetics allow for both systemic and direct urinary system action, as approximately 60% of an intravenously administered dose is excreted unchanged in urine.

While dedicated clinical trials focused on beta agonists for renal colic pain relief are lacking, a substantial body of evidence lends credence to their potential efficacy. This intriguing prospect warrants further exploration through rigorous research endeavors. Given the existing foundation of evidence, a systematic investigation into this treatment paradigm is a logical progression. Many studies have looked at treatments that might expedite stone passage. While this isn't the main focus of this trial, it is one of the secondary goals as previous research suggest salbutamol role in uteral relaxation.

Salbutamol's rapid onset of action, occurring within minutes, renders it an attractive option for addressing the sudden and severe pain characteristic of renal colic in the ED setting. Familiarity among emergency department staff further enhances its appeal, ensuring ease of administration. In this study, we propose a 10 mg nebulized salbutamol dose, an approved dosage that achieves systemic absorption, ensuring a therapeutic effect. Furthermore, this dosage is unlikely to exert undue influence on electrolyte balance and adheres to established guidelines for managing elevated blood potassium levels.

Considering safety, salbutamol's side effect profile, characterized by mild effects such as increased heart rate and shivering, is well-documented and understood, particularly when compared with alternative analgesics. Notably, salbutamol exhibits a relatively modest impact on blood potassium levels (lowering potassium level) compared to other analogous medications. However, studies have revealed that any potential potassium level alterations are primarily observed in individuals who are regular users of salbutamol, with no substantive changes noted in blood potassium levels in research involving salbutamol use, especially at doses ranging from 5mg to 10mg.

The scientific rationale underpinning the consideration of beta-agonists, like salbutamol, for renal colic pain relief rests upon their ability to ameliorate ureteral spasms, a principal contributor to the affliction of pain, subsequently abating the associated agony. Support for this hypothesis stems from an extensive body of evidence encompassing laboratory studies, animal experiments, and human investigations. Studies in human subjects have corroborated the premise that agents inducing ureteral relaxation can mitigate pain and potentially reduce the need for additional analgesic interventions.

In summary, the utilization of salbutamol as a potential therapeutic agent for renal colic pain relief represents an exciting frontier in medical research, offering a multifaceted approach to pain management. Its rapid onset, established safety profile, and plausible mechanistic underpinnings position it as a compelling candidate for further exploration and investigation. By embarking on this research journey, we aim to enhance our understanding of effective renal colic pain relief strategies and, in turn, advance patient care in this challenging clinical context.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with classical acute renal colic symptoms.
2. Age ≥ 18 years and < 60 years
3. Hemodynamically stable vital signs.
4. Mentally competent patient who can understand and sign the consent form.

Exclusion Criteria:

1. Patients who are allergic to Salbuamtol.
2. Renal disease or transplant.
3. Patients with pervious myocardial infarction and PCI.
4. Active peptic ulcer disease.
5. Liver cirrhosis.
6. Couagulopathy.
7. History of asthma , urticaria, or other allergic-type reactions after taking NSAIDs.
8. Patient with any other contraindications to use of NSAIDs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain reduction at 60 minutes | 60 minutes
  The Analgesic effects of Nebulized Salbutamol on patient with renal colic as measured by Numerical rating scale (NRS).Minimum of Zero and Maximum of Ten in Number scale , in which zero will be least pain expiernced and Ten is the worse pain expiernced by the patient. Increasing Number from (zero to ten) meaning Wrosning of pain.

SECONDARY OUTCOMES:
Adverse Event/Side Effects | 60 mintues
  sides effects will be monitored during the study protocol period like (nausea , vomiting , dizziness )
Need of Rescue medications | 60 mintues
  rate of recuse medications (Opioids )
Pain reduction rate. | 15, 30, 45, 60 mintues
  The rate of pain reduction will be monitored during the 60 minutes at each 15-minute interval.
ED revisits | 48 hrs
  Patient will be followed up after 48 hrs by a follow-up call to document ED revisits.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Al Shamsi, MD, Study Director — Armed Forces Hospital, Oman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chauhan CK, Joshi MJ, Vaidya AD. Growth inhibition of struvite crystals in the presence of herbal extract Commiphora wightii. J Mater Sci Mater Med. 2009 Dec;20 Suppl 1:S85-92. doi: 10.1007/s10856-008-3489-z. Epub 2008 Jun 21. PMID 18568390
- [Background] Teichman JM. Clinical practice. Acute renal colic from ureteral calculus. N Engl J Med. 2004 Feb 12;350(7):684-93. doi: 10.1056/NEJMcp030813. No abstract available. PMID 14960744
- [Background] Holdgate A, Pollock T. Systematic review of the relative efficacy of non-steroidal anti-inflammatory drugs and opioids in the treatment of acute renal colic. BMJ. 2004 Jun 12;328(7453):1401. doi: 10.1136/bmj.38119.581991.55. Epub 2004 Jun 3. PMID 15178585
- [Background] Tabner AJ, Johnson GD, Fakis A, Surtees J, Lennon RI. beta-Adrenoreceptor agonists in the management of pain associated with renal colic: a systematic review. BMJ Open. 2016 Jun 20;6(6):e011315. doi: 10.1136/bmjopen-2016-011315. PMID 27324714
- [Background] Pickard R, Starr K, MacLennan G, Lam T, Thomas R, Burr J, McPherson G, McDonald A, Anson K, N'Dow J, Burgess N, Clark T, Kilonzo M, Gillies K, Shearer K, Boachie C, Cameron S, Norrie J, McClinton S. Medical expulsive therapy in adults with ureteric colic: a multicentre, randomised, placebo-controlled trial. Lancet. 2015 Jul 25;386(9991):341-9. doi: 10.1016/S0140-6736(15)60933-3. Epub 2015 May 18. PMID 25998582
- [Background] Wanajo I, Tomiyama Y, Yamazaki Y, Kojima M. Ureteral selectivity of intravenous beta-adrenoceptor agonists in pig model of acute ureteral obstruction: comparison of KUL-7211, a selective beta2/beta3 agonist, with isoproterenol, terbutaline, and CL-316243. Urology. 2011 May;77(5):1266.e1-6. doi: 10.1016/j.urology.2010.12.045. Epub 2011 Mar 12. PMID 21397304
- [Background] Tomiyama Y, Murakami M, Hayakawa K, Akiyama K, Yamazaki Y, Kojima M, Shibata N, Akahane M. Pharmacological profile of KUL-7211, a selective beta-adrenoceptor agonist, in isolated ureteral smooth muscle. J Pharmacol Sci. 2003 Aug;92(4):411-9. doi: 10.1254/jphs.92.411. PMID 12939526